CLINICAL TRIAL: NCT05603910
Title: Phase 1 Clinical Trial of Lenvatinib, Pembrolizumab and Hypofractionated Pelvic Radiation Therapy for Mismatch Repair Proficient (pMMR) Recurrent/Unresectable Endometrial Carcinoma
Brief Title: Phase 1 Clinical Trial of Lenvatinib, Pembrolizumab and Hypofractionated Pelvic Radiation Therapy for pMMR Recurrent/Unresectable Endometrial Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aaron Wolfson (Other)
Responsible Party: Sponsor-Investigator, Aaron Wolfson, Professor of Radiation Oncology, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220813
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Endometrial Carcinoma; Unresectable Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lenvatinib, Pembrolizumab and Hypofractionated (Hypofx) External Beam Radiation Therapy (EBRT) Group (Experimental): Participants in this group will receive a combination treatment of Lenvatinib, Pembrolizumab, and Hypofx Pelvic EBRT over a period of approximately 10 to 12 weeks.
  1. Lenvatinib - administered in a 3 plus 3 escalation/de-escalation design. Participants will receive 1 of 4 of the following dose levels:
     Dose level 1- 4 mg Dose level 2- 8 mg Dose level 3 (Starting dose) - 12 mg Dose level 4- 16 mg
  2. Pembrolizumab- 200 mg IV will be administered on Day 1, 22 and 43
  3. HypoFx whole pelvic EBRT begins on Day 22 and continues for a total of 16 fractions of radiation given at a dose of 2.5 Gy per fraction for a total dose of 40.0 Gy delivered to the pelvis. A pelvic boost HypoFx EBRT consisting of 7 fractions of radiation given at a dose of 2.5 Gy per fraction that will be delivered to site(s) of gross disease of at least 1.0 cm in size. An additional boost total dose of 17.5 Gy administered will be administered over a period of 1.5 to 2.0 weeks.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab; Radiation: Hypofractionated External Beam Radiation Therapy

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsules taken daily by mouth
  Other Names: Lenvima
Drug: Pembrolizumab — 200 mg Pembrolizumab administered intravenously (IV) once on Days 1, 22 and 43.
  Other Names: Keytruda
Radiation: Hypofractionated External Beam Radiation Therapy — HypoFx whole pelvic EBRT begins on Day 22 and continues for a total of 16 fractions of radiation given at a dose of 2.5 Gy per fraction for a total dose of 40.0 Gy delivered to the pelvis. A pelvic boost HypoFx EBRT consisting of 7 fractions of radiation given at a dose of 2.5 Gy per fraction that will be delivered to site(s) of gross disease of at least 1.0 cm in size. An additional boost total dose of 17.5 Gy administered will be administered over a period of 1.5 to 2.0 weeks.

SUMMARY:
The purpose of this research study is to see if it is feasible to combine a fixed dose of pembrolizumab and a daily dose of oral lenvatinib, along with daily treatments of an abbreviated course of pelvic external beam radiation therapy, to support cancer cells in multiplying and spreading to other body sites.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven recurrent pMMR EC following surgery alone or de novo unresectable pMMR EC for whom External beam radiation therapy (EBRT) has been determined as an appropriate therapeutic approach. Eligible tumor histologies include the following: endometrioid adenocarcinoma, adenocarcinoma with squamous differentiation, mucinous, mixed carcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, and serous adenocarcinoma histologies as determined by tissue from an archival sample or newly obtained core or excisional biopsy of a tumor lesion. For patients with recurrent disease greater than six months (>6 months), a fresh biopsy must be obtained.
2. Measurable disease of at least 1.0 cm in size defined by RECIST 1.1 on imaging studies with at least one (1) site located in the pelvis and/or vagina without any foci of extra-pelvic disease (including the para-aortic region or inguinal-femoral lymph nodes).13
3. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Karnofsky score ≥50). See APPENDIX A.
4. Patients must have pMMR tumor subtype(s).
5. Patients must have normal organ and marrow function as defined below:

   System Laboratory Value Hematological Absolute neutrophil count (ANC)
   * 1,500 cells/mm³ Platelets
   * 100,000 cells/mm³ Hemoglobin
   * 9.0 g/dL Renal Serum creatinine or Measured or calculated a creatinine clearance glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)

     ≤ 1.5 x upper limit of normal (ULN) or CrCl ≥ 40 mL/min Hepatic Serum total bilirubin <1.0 ULN Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine transaminase (ALT) serum glutamic-pyruvic transaminase (SGPT) Aminotransferase (AST and ALT) ≤ 2.5 x ULN or 5 X ULN for patients with liver metastases Albumin
   * 2.5 mg/dL a CrCl should be calculated per institutional standard.
6. Female participants of childbearing potential (those who have not been surgically sterilized or have not been without menses for >1 year) should be willing to use 2 methods of birth control at the same time or be surgically sterile or abstain from heterosexual activity for the course of the study and for at least 120 days after the last study dose. For more information, see Section 4.8.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Women age ≥18 years old.

Exclusion Criteria:

1. Patients who are currently in or have participated in a study of an investigational agent or used an investigational device within 4 weeks of the first dose of study treatment.
2. Patients with Mismatch repair deficient (dMMR) and endometrial carcinomas.
3. Patients with dMMR and uterine carcinosarcomas.
4. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   EXCEPTION: Patients with previously treated brain metastases, including receiving prior brain irradiation, may participate provided they are stable (without evidence of progression by imaging for at least 3 months prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, are not using steroids for at least 28 days prior to study treatment, and have not received prior cranial irradiation for at least 3 months prior to study treatment.
5. Patients with a known additional malignancy that is progressing or requires active treatment.

   EXCEPTIONS include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Prior treatment with lenvatinib, anti-programmed cell death-1(PD)-1, anti-PD-L1, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
7. Patients who are planned to receive vaginal brachytherapy as their pelvic boost course of radiation as determined by their treating physician(s).
8. No prior radiation therapy to the vagina, pelvis, or abdomen will be allowed.
9. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or other serious medical condition or social situations that in the judgement of the Investigator(s) would interfere or limit compliance with study requirements/treatments.
10. Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 21 days prior to the first dose of study treatment.

    Note: Patients with active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs) and/or requiring replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. Evidence of uncontrolled hypertension as documented in the patient's medical record.
13. Known psychiatric illness/condition or substance abuse disorders that in the judgement of the Investigator(s) would interfere with cooperation with requirements of the study.
14. Is pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
15. Patients with uncontrolled human immunodeficiency virus (HIV) infection, which is defined as follows:

    1. Antiviral therapy treatment for <4 weeks AND
    2. Have an HIV viral load ≥400 copies/mL prior to enrollment.
16. Patients with uncontrolled hepatitis B virus (HBV) infection or who are chronic carriers of hepatitis B infection, which is defined as:

    1. Hepatitis B surface antigen reactive (HbsAg-positive), undetectable or low HBV DNA, and with normal ALT levels who are not on HBV therapy
    2. Individuals who have serologic evidence of a resolved prior HBV infection (ie, HBSAg-negative and anti-core hepatitis B antibody positive (anti-Hepatitis B core -positive)
17. Patients with active, untreated hepatitis C virus (HCV) infection or who have not completed their HCV antiviral regimen. Patients with a history of HCV infection may participate in this study if their HCV ribonucleic acid (RNA) level is below the limit of quantification.
18. Received live vaccine within 30 days prior to the first dose of study treatment.
19. Patient has active Mycobacterium tuberculosis infection (tuberculosis or TB).
20. A QT interval corrected for heart rate using Bazett's formula (QTcB) ≥ 480msec.
21. Patient receiving concurrent additional biologic therapy.
22. Patients with impaired decision-making capacity.
23. Patients who have not recovered from major surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of Lenvatinib | Up to 1 year
  The RP2D will be the highest dose of Lenvatinib that in combination with Pembrolizumab and Hypofractionated (HypoFx) pelvic External Beam Radiotherapy (EBRT) yields less than 2 Dose Limiting Toxicities (DLTs) in 6 patients.
Number of Events of Treatment-Related Toxicity | Up to 12 weeks
  The number of events of any treatment related (an attribution of definite, possible or probable relation to study treatment) DLTs and any toxicity or Adverse Events (AE) will be assessed by treating physician using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 weeks
  ORR is defined as the proportion of study patients achieving a Complete Response (CR) or Partial Response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Number of Reported Adverse Events | Up to 12 weeks
  All other reported adverse events regardless of physicians' assessment of relation to study drugs using NCI CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H Wolfson, MD, FACR, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No